CLINICAL TRIAL: NCT02914080
Title: Validation of a Psychological Fragility Questionnary in the Elderly in Isolation
Acronym: MUTAC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 14-PP-09
Record Dates: First submitted 2016-09-13; First posted 2016-09-26 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Loneliness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Social isolation and loneliness of the elderly have become major public health problems, because of the deleterious consequences if not lethal they can generate.

Because of frequent resignation to these phenomena, support must be given to all means of prevention to prevent or at least mitigate their impacts. It appears from the literature that are isolated or living as they have adjustment difficulties which are linked to fragility. If geriatric frailty have been defined to date in somatic and cognitive criteria, psychological fragility criteria have been little discussed outside of psychiatric disorders (depression, anxiety disorders in particular).

This study aims to test in the elderly in isolation psychological fragility questionnaire and to study the statistical qualities and relations with socio-demographic variables, environmental and other known vulnerabilities.

ELIGIBILITY:
Inclusion Criteria:

* People over 65
* Living alone at home (rural and urban ) or institution ( nursing home , no family member or spouse in the same institution).
* No not refusing to participate in the survey

Exclusion Criteria:

* Overt or decompensated psychiatric pathology: major depressive disorder , bipolar disorder, psychotic disorder, severe personality disorder , primary addiction ( ICD-10 criteria)
* Alzheimer's disease or related illness probable or confirmed (ICD criteria 10)
* Sequel to severe neurological disease , unstabilized somatic pathology and / or may disrupt data collection
* Patients do not have the capacity to understand the objectives of the survey

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly people living in isolation , will be tested in different environments : ( i) in rural areas; ( Ii ) in urban areas ; ( Iii) accommodation facility for elderly dependents ( EHPAD)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Psychological scales used to evaluate the elements of fragility in the elderly in isolation | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No